CLINICAL TRIAL: NCT00554606
Title: A 54-week, Phase II, Multi-center, Open-label Extension Study to Evaluate the Efficacy, Safety and Tolerability of ACZ885 (Anti-interleukin-1B Monoclonal Antibody) in Patients With Rheumatoid Arthritis
Brief Title: Long-term Efficacy, Safety and Tolerability of ACZ885 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885A2211
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anti-interleukin-1 beta; ACZ885
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canakinumab (Experimental): Participants received one single dose of 600 mg canakinumab via intravenous infusion on Day 1 and thereafter every 6 weeks until completion of the 54-week treatment period.
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — Canakinumab
  Other Names: ACZ885

SUMMARY:
This study will assess the long-term safety and tolerability of ACZ885 in patients with rheumatoid arthritis, as well as long-term efficacy, long-term preservation and/or improvement of joint structure and bone mineral density, and long term maintenance of health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and non-pregnant, non-lactating females) who completed the core CACZ885A2204, CACZ885A2206, or CACZ885A2207 study without serious or severe drug-related adverse effects may enter the extension study upon signing informed consent

Exclusion Criteria:

* Patients for whom continued treatment in the extension is not considered appropriate by the treating physician.
* Patients who were non-compliant or who demonstrated a major protocol violation in the core study.
* Patients who did not complete / discontinued from the core study.
* Patients with drug related serious adverse events or severe adverse events.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-10-11 (Actual); Primary Completion 2009-08-13 (Actual); Study Completion 2009-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (51):
- United States (20):
  - Novartis Investigator Site, Huntsville, Alabama
  - Novartis Investigator Site, Tuscaloosa, Alabama
  - Novartis Investigator Site, Paradise Valley, Arizona
  - Novartis Investigator Site, Trumbull, Connecticut
  - Novartis Investigator Site, Jacksonville, Florida
  - Novartis Investigator Site, South Miami, Florida
  - Novartis Investigator Site, Tamarac, Florida
  - Novartis Investigator Site, Rockford, Illinois
  - Novartis Investigator Site, Urbandale, Indiana
  - Novartis Investigator Site, Richmond Heights, Missouri
  - Novartis Investigator Site, Omaha, Nebraska
  - Novartis Investigator Site, Reno, Nevada
  - Novartis Investigator Site, Tulsa, Oklahoma
  - Novartis Investigator Site, Austin, Texas
  - Novartis Investigator Site, Carrollton, Texas
  - Novartis Investigator Site, Dallas, Texas
  - Novartis Investigator Site, Fort Worth, Texas
  - Novartis Investigator Site, Mesquite, Texas
  - Novartis Investigator Site, Arlington, Virginia
  - Novartis Investigator Site, Spokane, Washington
- Belgium (3):
  - Novartis Investigator Site, Antwerp
  - Novartis Investigator Site, Diepenbeek
  - Novartis Investigator Site, Liège
- Germany (6):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Ratingen
  - Novartis Investigator Site, Sendenhorst
  - Novartis Investigator Site, Wiesbaden
- Italy (4):
  - Novartis Investigator Site, Arenzano, GE
  - Novartis Investigator Site, Valeggio sul Mincio, VR
  - Novartis Investigator Site, Genova
  - Novartis Investigator Site, Padua
- Netherlands (3):
  - Novartis Investigator Site, Leeuwarden
  - Novartis Investigator Site, Leiden
  - Novartis Investigator Site, Venlo
- Russia (3):
  - Novartis Investigator Site, Moscow
  - Novartis Investigator Site, Yaroslavl
  - Novartis Investigator Site, Yekaterinburg
- Spain (7):
  - Novartis Investigator Site, Alicante
  - Novartis Investigator Site, Barcelona
  - Novartis Investigator Site, Bilbao
  - Novartis Investigator Site, Madrid
  - Novartis Investigator Site, Santiago de Compostela
  - Novartis Investigator Site, Seville
  - Novartis Investigator Site, Valencia
- Switzerland (2):
  - Novartis Investigator Site, Basel
  - Novartis Investigator Site, Zurich
- Turkey (Türkiye) (3):
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Izmir
  - Novartis Investigator Site, Sihhiye/Ankara

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 115 participants were enrolled in the trial (56 from core trial CACZ885A2204, 8 from CACZ885A2206, and 51 from CACZ885A2207).
Groups:
- Canakinumab (ACZ885): Participants received one single dose of 600 mg canakinumab via intravenous infusion on Day 1 and thereafter every 6 weeks until completion of the 54-week treatment period.
Period: Overall Study
Arm/Group | Canakinumab (ACZ885)
Started | 115
Completed | 30
Not Completed | 85
Not completed — Adverse Event | 3
Not completed — Abnormal laboratory values | 1
Not completed — Unsatisfactory therapeutic effect | 14
Not completed — Subject withdrew consent | 2
Not completed — Lost to Follow-up | 2
Not completed — Administrative problems | 60
Not completed — Death | 1
Not completed — Protocol deviation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
Age, Customized [Mean (Standard Deviation); unit: years] | 52.3 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 109
  Black | 2
  Asian | 2
  Native American | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: From start of the study up to End Of Study (Week 60)
Population: The Safety Analysis Set was defined as all participants that received at least one dose of study drug (in this extension) with at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
Participants
  Adverse Events | 91
  Death | 1
  Serious Adverse Events | 8
  Discontinued due to Serious Adverse Events | 3

2. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology Response 20 (ACR20)
Description: ACR20 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
percentage of participants
  Baseline | 48.7
  Day 1 | 49.6
  Week 6: number analyzed (Participants) | 108
  Week 6 | 57.4
  Week 12: number analyzed (Participants) | 107
  Week 12 | 53.3
  Week 18: number analyzed (Participants) | 104
  Week 18 | 58.7
  Week 24: number analyzed (Participants) | 96
  Week 24 | 54.2
  Week 30: number analyzed (Participants) | 83
  Week 30 | 61.4
  WeeK 36: number analyzed (Participants) | 74
  WeeK 36 | 52.7
  Week 42: number analyzed (Participants) | 49
  Week 42 | 57.1
  Week 48: number analyzed (Participants) | 45
  Week 48 | 53.3
  Week 54 (Follow-Up): number analyzed (Participants) | 48
  Week 54 (Follow-Up) | 41.7
  End of Study: number analyzed (Participants) | 111
  End of Study | 45.9

3. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology Response 50 (ACR50)
Description: ACR50 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 50% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
percentage of participants
  Baseline | 23.5
  Day 1 | 23.5
  Week 6: number analyzed (Participants) | 108
  Week 6 | 25.0
  Week 12: number analyzed (Participants) | 107
  Week 12 | 30.8
  Week 18: number analyzed (Participants) | 104
  Week 18 | 26.0
  Week 24: number analyzed (Participants) | 96
  Week 24 | 32.3
  Week 30: number analyzed (Participants) | 83
  Week 30 | 32.5
  Week 36: number analyzed (Participants) | 74
  Week 36 | 35.1
  Week 42: number analyzed (Participants) | 49
  Week 42 | 38.8
  Week 48: number analyzed (Participants) | 45
  Week 48 | 28.9
  End of Study: number analyzed (Participants) | 111
  End of Study | 26.1

4. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology Response 70 (ACR70)
Description: ACR70 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 70% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
percentage of participants
  Baseline | 12.2
  Day 1 | 11.3
  Week 6: number analyzed (Participants) | 108
  Week 6 | 13.0
  Week 12: number analyzed (Participants) | 107
  Week 12 | 13.1
  Week 18: number analyzed (Participants) | 104
  Week 18 | 14.4
  Week 24: number analyzed (Participants) | 96
  Week 24 | 16.7
  Week 30: number analyzed (Participants) | 83
  Week 30 | 18.1
  Week 36: number analyzed (Participants) | 74
  Week 36 | 20.3
  Week 42: number analyzed (Participants) | 49
  Week 42 | 26.5
  Week 48: number analyzed (Participants) | 45
  Week 48 | 13.3
  Week 54 (Follow-Up): number analyzed (Participants) | 48
  Week 54 (Follow-Up) | 14.6
  End of Study: number analyzed (Participants) | 111
  End of Study | 15.3

5. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology Response 90 (ACR90)
Description: ACR90 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 90% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: The Safety Analysis Set was defined as all subjects that received at least one dose of study drug (in this extension) with at least one post-baseline safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
percentage of participants
  Baseline | 2.6
  Day 1 | 2.6
  Week 6: number analyzed (Participants) | 108
  Week 6 | 2.8
  Week 12: number analyzed (Participants) | 107
  Week 12 | 2.8
  Week 18: number analyzed (Participants) | 104
  Week 18 | 1.9
  Week 24: number analyzed (Participants) | 96
  Week 24 | 5.2
  Week 30: number analyzed (Participants) | 83
  Week 30 | 3.6
  Week 36: number analyzed (Participants) | 74
  Week 36 | 6.8
  Week 42: number analyzed (Participants) | 49
  Week 42 | 8.2
  Week 48: number analyzed (Participants) | 45
  Week 48 | 6.7
  Week 54 (Follow-Up): number analyzed (Participants) | 48
  Week 54 (Follow-Up) | 10.4
  End of Study: number analyzed (Participants) | 111
  End of Study | 5.4

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on Disease Activity Score (DAS) 28 and Simplified Disease Activity Index (SDAI)
Description: At each visit (including baseline) the DAS28 and SDAI variables were derived using the following formulas:
  DAS28 = 0.56*√ (tender28) + 0.28 * √ (swollen28) + 0.36 * loge(CRP+1) + 0.014*PGDA+ 0.96; SDAI = tender28 + swollen28 + CRP + (PGDA / 10) + (EGDA / 10) where tender28 is the tender 28-joint count, swollen28 is the swollen 28-joint count, CRP is C-reactive protein, PGDA is the patient's global assessment of disease activity and EGDA is the physician's global assessment of disease activity.
  The Number of Participants in clinical remission is defined as the DAS28 ≤ (less than or equal to) 2.6 or SDAI ≤ (less than or equal to) to3.3.
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
percentage of participants
  Baseline | 11.3
  Day 1 | 14.8
  Week 6: number analyzed (Participants) | 108
  Week 6 | 16.7
  Week 12: number analyzed (Participants) | 107
  Week 12 | 18.7
  Week 18: number analyzed (Participants) | 104
  Week 18 | 19.2
  Week 24: number analyzed (Participants) | 96
  Week 24 | 20.8
  Week 30: number analyzed (Participants) | 83
  Week 30 | 24.1
  Week 36: number analyzed (Participants) | 74
  Week 36 | 18.9
  Week 42: number analyzed (Participants) | 49
  Week 42 | 32.7
  Week 48: number analyzed (Participants) | 45
  Week 48 | 17.8
  Week 54 (Follow-Up): number analyzed (Participants) | 47
  Week 54 (Follow-Up) | 27.7
  End of study: number analyzed (Participants) | 110
  End of study | 18.2

7. Secondary Outcome: Change From Baseline in ACR Component : Swollen Joint Count Through Week 54
Description: Synovial fluid and/or soft tissue swelling but not bony overgrowth represents a positive result for swollen joint count. Joint counts were performed according to the visit schedule by the physician or by well trained personnel. Whenever possible, the same evaluator performed these assessments at all visits. The following 28 joints were assessed for tenderness and swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). If the number of joints for which data were available (e.g., S) was less than 28, the number of swollen joints (e.g., s) was scaled up proportionately (i.e., 28*(s/S)).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
Joints
  Baseline | 6.0 (5.10)
  Day 1 | 6.5 (5.53)
  Week 6 | 5.8 (5.65)
  Week 12 | 5.2 (5.16)
  Week 18 | 5.0 (5.18)
  Week 24 | 4.4 (4.35)
  Week 30 | 3.9 (4.37)
  Week 36 | 3.5 (4.65)
  Week 42 | 3.8 (4.60)
  Week 48 | 4.4 (4.99)
  Week 54 (Follow-Up) | 3.9 (5.22)
  End of Study | 5.1 (5.18)

8. Secondary Outcome: Change From Baseline in ACR Component : Tender Joint Count Through Week 54
Description: The ACR tender joint count (28 joints) was done by scoring several different aspects of tenderness as assessed by pressure and joint manipulation on physical examination. Joint counts were performed according to the visit schedule by the physician or by well trained personnel. The following 28 joints were assessed for tenderness and swelling: metacarpophalangeal I-V (10), thumb interphalangeal (2), hand proximal interphalangeal II-V (8), wrist (2), elbow (2), shoulders (2), and knees (2). If the number of joints for which data were available (e.g., T) was less than 28, the number of tender joints (e.g., t) was scaled up proportionately (i.e., 28*(t/T)).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
Joints
  Baseline | 9.3 (7.70)
  Day 1 | 9.5 (8.11)
  Week 6 | 8.7 (7.70)
  Week 12 | 7.9 (7.17)
  Week 18 | 7.7 (7.15)
  Week 24 | 7.1 (7.40)
  Week 30 | 6.9 (7.54)
  Week 36 | 6.9 (7.19)
  Week 42 | 3.8 (6.12)
  Week 48 | 4.9 (6.33)
  Week 54 (Follow-Up) | 5.9 (7.11)
  End of Study | 7.6 (7.25)

9. Secondary Outcome: Change From Baseline in ACR Component: Patient's Assessment of Pain Activity Through Week 54
Description: ACR components included patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimetres
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
millimetres
  Baseline | 42.3 (21.93)
  Day 1 | 41.2 (21.60)
  Week 6 | 37.8 (21.16)
  Week 12 | 37.1 (21.21)
  Week 18 | 39.4 (21.35)
  Week 24 | 36.8 (20.55)
  Week 30 | 36.3 (21.13)
  Week 36 | 36.5 (23.01)
  Week 42 | 32.5 (21.11)
  Week 48 | 33.0 (21.24)
  Week 54 (Follow-Up) | 35.9 (22.12)
  End of Study | 40.1 (20.60)

10. Secondary Outcome: Change From Baseline in ACR Component:- Patient's Global Assessment of Disease Activity Through Week 24
Description: ACR component included patient's global assessment (PtGA) of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
millimeters
  Baseline | 45.0 (23.05)
  Day 1 | 44.1 (21.96)
  Week 6 | 40.3 (22.02)
  Week 12 | 39.9 (21.01)
  Week 18 | 42.0 (20.89)
  Week 24 | 38.3 (21.04)
  Week 30 | 36.6 (21.97)
  Week 36 | 39.9 (21.70)
  Week 42 | 31.2 (21.40)
  Week 48 | 37.6 (23.08)
  Week 54 (Follow-Up) | 38.4 (23.99)
  End of Study | 42.0 (21.77)

11. Secondary Outcome: Change From Baseline in ACR Component : Physician's Global Assessment of Disease Activity Through Week 54
Description: ACR component included physician's global assessment (PGA) of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
millimeters
  Baseline | 37.0 (23.11)
  Day 1 | 38.7 (23.09)
  Week 6 | 34.1 (22.70)
  Week 12 | 33.0 (21.82)
  Week 18 | 33.7 (22.06)
  Week 24 | 27.8 (20.25)
  Week 30 | 26.0 (16.79)
  Week 36 | 24.6 (16.35)
  Week 42 | 21.3 (17.25)
  Week 48 | 23.3 (18.10)
  Week 54 (Follow-Up) | 27.6 (23.70)
  End of Study | 32.7 (22.88)

12. Secondary Outcome: Change From Baseline in ACR Component : C-reactive Protein (CRP) Through Week 54
Description: Blood for this assessment was obtained in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment. Assessment was performed by the central laboratory.
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams/liter
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
milligrams/liter
  Baseline: number analyzed (Participants) | 99
  Baseline | 14.42 (22.406)
  Day 1: number analyzed (Participants) | 114
  Day 1 | 15.30 (26.827)
  Week 6: number analyzed (Participants) | 108
  Week 6 | 10.38 (16.717)
  Week 12: number analyzed (Participants) | 105
  Week 12 | 10.10 (19.355)
  Week 18: number analyzed (Participants) | 101
  Week 18 | 9.99 (16.948)
  Week 24: number analyzed (Participants) | 89
  Week 24 | 8.35 (16.413)
  Week 30: number analyzed (Participants) | 75
  Week 30 | 8.03 (14.065)
  Week 36: number analyzed (Participants) | 62
  Week 36 | 6.49 (10.146)
  Week 42: number analyzed (Participants) | 35
  Week 42 | 5.71 (10.577)
  Week 48: number analyzed (Participants) | 33
  Week 48 | 6.72 (11.545)
  Week 54 (Follow-Up): number analyzed (Participants) | 35
  Week 54 (Follow-Up) | 6.71 (12.611)
  End of Study: number analyzed (Participants) | 106
  End of Study | 10.74 (22.520)

13. Secondary Outcome: Core Study Change From Baseline in Edema, Erosion and Synovitis Score Was Assessed at Week 18
Description: The MRI scan was scored according to OMERACT RAMRIS system. Erosions were scored on a scale of 0-10 per site, the scale is 0-10, based on the proportion of eroded bone compared to the "assessed bone volume", judged on all available images-0: no erosion; 1: 1-10% of bone eroded; 2; 11-20%, etc. For long bones, the "assessed bone volume" is from the articular surface (or its best estimated position if absent) to a depth of 1 cm, and in carpal bones it is the whole bone.
  Edema were scored on a scale of 0-10 per site, the scale is 0-3 based on the proportion of bone with edema, as follows-0: no edema; 1: 1-33% of bone edematous; 2: 34-66% of bone edematous; 3: 67-100%; and Synovitis on a scale of 0-3 per site, the scale is 0-3. Score 0 is normal, and 1-3 (mild, moderate, severe) are by thirds of the presumed maximum volume of enhancing tissue in the synovial compartment.
Time Frame: Baseline, Week 18
Population: The Safety Analysis Set was defined as all participants that received at least one dose of study drug. Here, number of participants (N) analyzed included all participants who were evaluable for this outcome measure and number analyzed (n) included all participants who were evaluable for the specified categories.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Canakinumab (ACZ885) (Core Trial CACZ885A2204): Participants received one single dose of 600 mg canakinumab via intravenous infusion on Day 1, 15 continuing every 4 weeks up to week 26 in the core trial CACZ885A2204.
- Non- ACZ885 ( (Core Trial CACZ885A2204)): Participant who did not receive ACZ885 (Canakinumab) in the core trial CACZ885A2204.
Arm/Group | Canakinumab (ACZ885) (Core Trial CACZ885A2204) | Non- ACZ885 ( (Core Trial CACZ885A2204))
Number analyzed (Participants) | 32 | 15
score on a scale
  Edema Score: number analyzed (Participants) | 26 | 14
  Edema Score | 0 [-0.39 to 0.04] | -0.043 [-0.86 to 3.00]
  Erosion Score | 0 [-0.13 to 0.09] | 0 [-0.39 to 0.30]
  Synovitis Score: number analyzed (Participants) | 27 | 11
  Synovitis Score | -0.143 [-1.86 to 0.57] | -0.714 [-1.43 to 0.14]

14. Secondary Outcome: Core Study Change From Baseline in Van Der Heijde Modified Total Sharp Score Was Assessed for Erosion Score at Week 18
Description: Digital radiographic (X-ray) assessment of 16 joints and bones in the hand and wrist were assessed for and 15 joints in the hand and wrist were assessed for joint space narrowing. Scoring of the radiographic assessment was according to modified Sharp/van der Heijde score. The maximum number of erosions is 160 in the hands and 120 in the feet; and the maximum scores for joint space narrowing are 120 and 48, respectively. Erosions are scored 1 for a discrete interruption of the cortical surface, and scored 2-5 for a larger defect according to the surface area of the joint involved. Notably, the maximum erosion score in each joint in hands is 5, while it is 10 in the feet. For joint space narrowing, 0=normal; 1=focal or doubtful; 2=general, <50% of the original joint space; 3=general, >50% of the original joint space or subluxation; 4=ankylosis.
Time Frame: Baseline, Week 18
Population: The Safety Analysis Set was defined as all participants that received at least one dose of study drug. Here, number of participants analyzed (N) included all participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Canakinumab (ACZ885) (Core Trial CACZ885A2204) | Non- ACZ885 ( (Core Trial CACZ885A2204))
Number analyzed (Participants) | 33 | 16
score on a scale
  Left Hand | 0 [-0.06 to 0.13] | 0 [0.00 to 0.63]
  Right Hand | 0 [0.00 to 0.25] | 0 [0.00 to 0.38]
  Left Foot | 0 [-0.17 to 1.00] | 0 [0.00 to 0.50]
  Right Foot | 0 [0.00 to 1.00] | 0 [0.00 to 0.67]

15. Secondary Outcome: Core Study Change From Baseline in Van Der Heijde Modified Total Sharp Score Was Assessed for Joint Narrowing Score at Week 18
Description: as for outcome 14
Time Frame: Baseline, Week 18
Population: The Safety Analysis Set was defined as all participants that received at least one dose of study drug (in this extension) with at least one post-baseline safety assessment. Here, N (number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Canakinumab (ACZ885) (Core Trial CACZ885A2204) | Non- ACZ885 ( (Core Trial CACZ885A2204))
Number analyzed (Participants) | 33 | 16
score on a scale
  Left Hand | 0 [0.00 to 0.13] | 0 [-0.07 to 0.07]
  Right Hand | 0 [-0.07 to 0.07] | 0 [-0.07 to 0.07]
  Left Foot | 0 [0.00 to 0.50] | 0 [0.00 to 0.00]
  Right Foot | 0 [0.00 to 0.17] | 0 [0.00 to 0.00]

16. Secondary Outcome: Core Study BMD of Total Lumbar Spine, Hip and Hand Was Assessed by DXA at Week 18
Description: Bone Mineral Density was measured by dual-energy X-ray absorptiometry (DXA) of the hand with the most swollen wrist (determined at baseline by the investigator site), lumbosacral (LS) spine and hip, in selected study sites. The reading of the DXA scans were performed centrally, by an experienced independent reader who was blinded to clinical details and MRI findings.
Time Frame: Baseline, Week 18
Population: The Safety Analysis Set was defined as all participants that received at least one dose of study drug. Number of participants analyzed signifies those who were evaluable for the assessment. Here, N (number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Canakinumab (ACZ885) (Core Trial CACZ885A2204) | Non- ACZ885 ( (Core Trial CACZ885A2204))
Number analyzed (Participants) | 4 | 1
g/cm2
  AP lumbar spine L1- L4 | 1.1650 (0.36399) | 1.1760
  Total Hip | 0.9000 (0.32558) | 0.8570
  Total Hand | 0.3295 (0.09726) | 0.4280

17. Secondary Outcome: Number of Subjects With Long-term Immunogenicity
Description: Anti-ACZ885 antibodies concentrations were assessed in serum. All blood samples were taken by direct venipuncture in a forearm vein. Immunogenicity was analyzed by BIAcore technology. immunogenicity was categorized as NO (no immunogenicity), BLQ (positive immunogenicity < LLOQ (not quantifiable)), and ALQ (positive immunogenicity > LLOQ (quantifiable).
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
Participants
  Baseline - No immunogenicity | 108
  Baseline - BLQ | 0
  Baseline - ALQ | 1
  DAY 1 - No immunogenicity | 94
  DAY 1 - BLQ | 0
  DAY 1 - ALQ | 0
  WEEK 6 - No immunogenicity | 1
  WEEK 6 - BLQ | 0
  WEEK 6 - ALQ | 0
  WEEK 12 - No immunogenicity | 89
  WEEK 12 - BLQ | 0
  WEEK 12 - ALQ | 0
  WEEK 24 - No immunogenicity | 73
  WEEK 24 - BLQ | 0
  WEEK 24 - ALQ | 0
  WEEK 36 - No immunogenicity | 46
  WEEK 36 - BLQ | 0
  WEEK 36 - ALQ | 0
  WEEK 48 - No immunogenicity | 21
  WEEK 48 - BLQ | 0
  WEEK 48 - ALQ | 0
  End of study - No immunogenicity | 93
  End of study - BLQ | 0
  End of study - ALQ | 0

18. Secondary Outcome: Pharmacokinetic (PK) of ACZ885: Systemic Clearance From Serum Following Intravenous Administration (CL) in Participants
Description: The PK parameter were evaluated from serum concentration-time data using mixed effects modeling approach.
Time Frame: Pre dose at Day 1, Pre dose at week 6, 12, 18, 24, 30, 36, 42, 48, follow up and at study completion (week 60)
Population: The PK set consisted of all participant who received at least one dose of study drug (in this extension) with at least one post-baseline pharmacokinetic assessment.
Measure: Mean (Standard Deviation); unit: Litre/day (L/d)
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
Litre/day (L/d) | 0.210 (0.0741)

19. Secondary Outcome: Pharmacokinetic (PK) of ACZ885: Volume Distribution From Serum Following Intravenous Administration (CL) in Participants
Description: The PK parameter were evaluated from serum concentration-time data using mixed effects modeling approach.
Time Frame: Pre dose at Day 1, Pre dose at week 6, 12, 18, 24, 30, 36, 42, 48, follow up and at study completion (week 60)
Population: The PK set consisted of all participants who received at least one dose of study drug (in this extension) with at least one post-baseline pharmacokinetic assessment.
Measure: Mean (Standard Deviation); unit: Litre (L)
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
Litre (L) | 3.34 (1.03)

20. Secondary Outcome: Health-Related Quality of Life (HRQoL) Accessed by Short Form (SF) -36 Score (Physical Component)
Description: The SF-36 measures the impact of disease on overall quality of life and consists of eight subscales (physical function, pain, general and mental health, vitality, social function, physical and emotional health) which can be aggregated to derive a physical-component summary score and a mental-component summary score.The scores range for each subscale from 0 to 10, and the composite score ranges from 0 to 100, with higher scores indicative of better health.
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: The safety population consisted of all randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
score on a scale
  Baseline: number analyzed (Participants) | 101
  Baseline | 38.115 (9.9799)
  Day 1: number analyzed (Participants) | 0
  Week 6: number analyzed (Participants) | 0
  Week 12: number analyzed (Participants) | 91
  Week 12 | 39.374 (9.7656)
  Week 18: number analyzed (Participants) | 0
  Week 24: number analyzed (Participants) | 81
  Week 24 | 39.437 (9.2349)
  Week 30: number analyzed (Participants) | 0
  Week 36: number analyzed (Participants) | 55
  Week 36 | 38.264 (10.0517)
  Week 42: number analyzed (Participants) | 0
  Week 48: number analyzed (Participants) | 30
  Week 48 | 40.110 (10.3660)
  Week 54 (Follow-Up): number analyzed (Participants) | 0
  End Of Study: number analyzed (Participants) | 103
  End Of Study | 38.295 (9.4491)

21. Secondary Outcome: Health-Related Quality of Life (HRQoL) Accessed by Health Assessment Questionnaire (HAQ) Score
Description: HAQ assesses the degree of difficulty experienced in 8 domains of daily living activities using 20 questions. The domains are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities, and each domain consists of 2 or 3 items. For each question, the level of difficulty is scored from 0 to 3 where 0 = without any difficulty (the best outcome), 1 = with some difficulty, 2 = much difficulty, and 3 = unable to do (the worst outcome). Each category is given a score by taking the maximum score of each question.A decrease from baseline indicates improvement for HAQ-DI. The HAQ-DI was calculated by dividing the sum of the category scores by the number of categories with at least 1 question answered. The HAQ-DI total score ranges from 0 to 3, with higher scores indicating greater disability.
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: The safety population consisted of all randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
units on a scale
  Baseline | 1.107 (0.6957)
  Day 1 | 1.039 (0.7271)
  Week 6 | 0.981 (0.6990)
  Week 12 | 1.044 (0.6924)
  Week 18 | 1.061 (0.7182)
  Week 24 | 0.997 (0.7224)
  Week 30 | 0.993 (0.7223)
  Week 36 | 1.008 (0.7450)
  Week 42 | 0.814 (0.8368)
  Week 48 | 0.837 (0.7529)
  Week 54 (Follow-Up) | 0.859 (0.7231)
  End of Study | 1.089 (0.7350)

22. Secondary Outcome: Health-Related Quality of Life (HRQoL) Accessed by Short Form (SF) -36 Score (Mental Component)
Description: as for outcome 20
Time Frame: Baseline Up to End Of Study (up to week 60)
Population: The safety population consisted of all randomized participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 115
score on a scale
  Baseline: number analyzed (Participants) | 101
  Baseline | 44.947 (11.9800)
  Day 1: number analyzed (Participants) | 0
  Week 6: number analyzed (Participants) | 0
  Week 12: number analyzed (Participants) | 91
  Week 12 | 45.867 (12.5364)
  Week 18: number analyzed (Participants) | 0
  Week 24: number analyzed (Participants) | 81
  Week 24 | 44.701 (11.9993)
  Week 30: number analyzed (Participants) | 0
  Week 36: number analyzed (Participants) | 55
  Week 36 | 45.175 (12.1436)
  Week 42: number analyzed (Participants) | 0
  Week 48: number analyzed (Participants) | 30
  Week 48 | 49.993 (13.0069)
  Week 54 (Follow-Up): number analyzed (Participants) | 0
  End Of Study: number analyzed (Participants) | 103
  End Of Study | 42.346 (11.8792)

ADVERSE EVENTS:
Time Frame: Adverse events were collected From Start of the Study up to EOS (Week 60)
Arm/Group | Canakinumab (ACZ885)
All-Cause Mortality (participants affected / at risk) | 1/115
Serious Adverse Events (participants affected / at risk) | 8/115
Other Adverse Events (participants affected / at risk) | 91/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=115)
Radius Fracture (Injury, poisoning and procedural complications) | 1
Lumbar Pain (Musculoskeletal and connective tissue disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Intermediate Uveitis (Eye disorders) | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1
Burn of internal organs (Injury, poisoning and procedural complications) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canakinumab (ACZ885) (N=115)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (6)
Odema peripheral (General disorders) | 4 (5)
Bronchitis (Infections and infestations) | 8 (9)
Gastroenteritis (Infections and infestations) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 7 (11)
Urinary tract infection (Infections and infestations) | 3 (4)
Blood pressure increased (Investigations) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Hepatic enzyme increased (Investigations) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (9)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 (9)
Headache (Nervous system disorders) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin reaction (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.